CLINICAL TRIAL: NCT04416165
Title: Comparison of FDG and FAPI in Patients With Various Types of Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019-XJS-1130
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Last update posted 2023-08-08 (Actual); Status verified 2023-06

CONDITIONS: Tumor, Solid; Positron-Emission Tomography; Metastasis
Keywords: Positron-Emission Tomography; Tumor, Solid; Diagnosis; Metastasis
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis; Disease

STUDY DESIGN:
Intervention Model Description: Subjects with various types of cancer undergo contemporaneous 68Ga-DOTA-FAPI-04 and 18F-FDG PET/CT either for an initial assessment or for recurrence detection.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental: 68Ga-DOTA-FAPI-04 (Experimental): Each subject receive a single intravenous injection of 18F-FDG and 68Ga-DOTA-FAPI-04, and undergo PET/CT imaging within the specified time.
  Interventions: Diagnostic Test: 18F-FDG and 68Ga-DOTA-FAPI -04 PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-FDG and 68Ga-DOTA-FAPI -04 PET/CT — Each subject receive a single intravenous injection of 18F-FDG and 68Ga-DOTA-FAPI-04, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the potential usefulness of 68Ga-DOTA-FAPI-04 positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various types of cancer, compared with 18F-FDG PET/CT.

DETAILED DESCRIPTION:
Subjects with various types of cancer underwent contemporaneous 68Ga-DOTA-FAPI-04 and 18F-FDG PET/CT either for an initial assessment or for recurrence detection. Tumor uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 68Ga-DOTA-FAPI-04 PET/CT were calculated and compared to evaluate the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order); (ii) patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report); (iii) patients who had scheduled both 18F-FDG and 68Ga-DOTA-FAPI-04 PET/CT scans; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions; (ii) patients with pregnancy; (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3000 (Estimated)
Dates: Start 2019-10-20 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
SUV | 30 days
  Standardized uptake value (SUV) of 18F/ 68Ga-DOTA-FAPI-04 for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-FDG and 68Ga-DOTA-FAPI-04 PET/CT were calculated and compared to evaluate the diagnostic efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- First affiliated hospital of xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo W, Pang Y, Yao L, Zhao L, Fan C, Ke J, Guo P, Hao B, Fu H, Xie C, Lin Q, Wu H, Sun L, Chen H. Imaging fibroblast activation protein in liver cancer: a single-center post hoc retrospective analysis to compare [68Ga]Ga-FAPI-04 PET/CT versus MRI and [18F]-FDG PET/CT. Eur J Nucl Med Mol Imaging. 2021 May;48(5):1604-1617. doi: 10.1007/s00259-020-05095-0. Epub 2020 Nov 11. PMID 33179149